CLINICAL TRIAL: NCT06327204
Title: Efficacy of Different Low Level Laser Therapy Sessions in Management of Masseter Muscle Trigger Points
Brief Title: Efficacy of Different Low Level Laser Therapy Sessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amany Ahmed AlAraby, lecturer of Oral Medicine, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Low Level laser 24
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Myofascial Pain Syndrome
Keywords: Trigger Point Pain, Myofascial, Laser therapy
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): patient received one session / week
  Interventions: Device: 940-nm diode laser / one session
- group II (Active Comparator): patient received two session / week
  Interventions: Device: 940-nm diode laser / two session
- Group III (Active Comparator): Patient received three session / week
  Interventions: Device: 940-nm diode laser/ three session

INTERVENTIONS:
Device: 940-nm diode laser / one session — laser therapy using a 940-nm diode laser / one session per week
  Arms: Group I
Device: 940-nm diode laser / two session — laser therapy using a 940-nm diode laser / two session per week
  Arms: group II
Device: 940-nm diode laser/ three session — laser therapy using a 940-nm diode laser / three session per week
  Arms: Group III

SUMMARY:
Myofascial pain dysfunction syndrome is one of the common causes of non-odontogenic pain in the head and neck region. It accounts for 40-60% of the adult population. Different treatment modalities had been reported to release the trigger point within the muscles of mastication in order to reduce pain and allow recovery of the function.

DETAILED DESCRIPTION:
Low-level laser therapy has been a research focus in past few years as it provides effective and conservative treatment modality with minimal patient discomfort. LLLT promotes the release of endogenous opioids, enhance tissue repair and cellular respiration, increase vasodilatation and pain relief Recent systematic review and meta-analysis had reported that the available evidence didn't allow clinicians to draw firm conclusions on effective dosage. This study aimed to investigate the effect of different LLLT sessions' number on pain, maximum mouth opening and quality of life in patients with masseter muscle trigger points.

ELIGIBILITY:
Inclusion Criteria:

1. definite diagnosis of myofascial pain based on the DC/TMD criteria with a referral
2. presence of one or more trigger points in the masseter muscle
3. no history of any invasive procedures of the related masseter muscle.

Exclusion Criteria:

1. any painful conditions affecting the orofacial region
2. any systemic diseases that could masticatory function (e.g., rheumatoid arthritis and epilepsy)
3. pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
pain score | 8 weeks
  a 10-point visual analogue score

SECONDARY OUTCOMES:
maximum mouth opening | 8 weeks
  measuring the interincisal distance between the upper and lower central incisors
quality of life questioner | 8 weeks
  Oral Health Impact Profile questionnaire (OHIP-14) containing 14 questions divided into seven domains of oral health

CONTACTS AND LOCATIONS:
Overall Officials: amany Ahmed, PhD, Principal Investigator — faculty of dentistry, October 6 University, Egypt
Locations (1):
- Faculty of Dentistry, October 6 University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahrari F, Madani AS, Ghafouri ZS, Tuner J. The efficacy of low-level laser therapy for the treatment of myogenous temporomandibular joint disorder. Lasers Med Sci. 2014 Mar;29(2):551-7. doi: 10.1007/s10103-012-1253-6. Epub 2013 Jan 15. PMID 23318917
- [Background] Maia ML, Bonjardim LR, Quintans Jde S, Ribeiro MA, Maia LG, Conti PC. Effect of low-level laser therapy on pain levels in patients with temporomandibular disorders: a systematic review. J Appl Oral Sci. 2012 Nov-Dec;20(6):594-602. doi: 10.1590/s1678-77572012000600002. PMID 23329239
- [Derived] Mahmoud NR, Shehab WI, AlAraby AA, Habaka YF. Efficacy of different low-level laser therapy sessions in the management of masseter muscle trigger points. BMC Oral Health. 2024 Sep 26;24(1):1125. doi: 10.1186/s12903-024-04780-y. PMID 39327563